CLINICAL TRIAL: NCT03755206
Title: Sust-AIns: Sustainment of Suicide Prevention Programs in American Indian Settings
Acronym: Sust-AIns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00008138
Record Dates: First submitted 2018-11-20; First posted 2018-11-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Program Sustainability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): Interrupted time series design
  Interventions: Other: Sustainability strategies

INTERVENTIONS:
Other: Sustainability strategies — The investigators will work with each site to determine strategies that are relevant locally to help promote sustainability of the suicide prevention program.

SUMMARY:
The proposed study is part of the research project for a National Institute of Mental Health K01 grant to Dr. Haroz. The overall research project is focused on understanding how to sustain evidenced-based mental and behavioral health programs in tribal contexts. The aim of this study is to pilot test sustainment strategy interventions across tribal settings using mixed-methods.

DETAILED DESCRIPTION:
Among the most pressing issues in mental health Dissemination and Implementation research (D&I) is the lack of knowledge about how to sustain mental health prevention and treatment services for which there is substantial evidence of impact. Most D&I studies focus on adoption and initial implementation, with few studies (<20) rigorously exploring sustainment. The sustainment of services has been described as "one of the greatest, yet least understood, challenges in the field of implementation science." The gap in knowledge is even greater for low-resource contexts, as few studies have focused on these settings. This project aims to address this gap by developing and testing sustainment strategies for an evidenced-based youth suicide prevention program in a low-resource, American Indian (AI) contexts.

ELIGIBILITY:
Inclusion Criteria:

* Knowledgeable about the implementation of the suicide prevention program
* Over the age of 18
* Available to participate in required study meetings and assessments
* Fluent in English

Exclusion Criteria:

* Factors identified at baseline that preclude full participation including: being under the influence of a substance; active psychosis or mania; any other condition that makes an individual lack capacity to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily E. Haroz, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Online Survey, Whiteriver, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- No Allocation: N/A No Allocation
  Sustainability strategies: The investigators will work with each site to determine strategies that are relevant locally to help promote sustainability of the suicide prevention program.
Arm/Group | No Allocation
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 24
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24
Program Sustainability Assessment Tool [Mean (Standard Deviation); unit: units on a scale] — Possible score range 0-3, higher scores indicate more capacity for program sustainability
  units on a scale | 2.2 (0.42)

OUTCOME MEASURES:

1. Primary Outcome: Program Sustainability Assessment Tool
Description: Tool that assess domains of capacity for sustainability. Possible score range 0-3, higher scores indicate more capacity for program sustainability.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sustainability Strategies
Number analyzed (Participants) | 24
score on a scale | 2.1 (0.53)

ADVERSE EVENTS:
Description: There were no adverse event tracking or reporting. It was declared non-human subjects research as it focused on understanding implementation.
Groups:
- Sustainability Strategies: Interrupted time series design
  Sustainability strategies: The investigators will work with each site to determine strategies that are relevant locally to help promote sustainability of the suicide prevention program.
Arm/Group | Sustainability Strategies
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT03755206/Prot_SAP_000.pdf